CLINICAL TRIAL: NCT03200600
Title: Impact of Perioperative Dexamethasone and Flurbiprofen Axetil on Delirium After Surgery for Non-small Cell Lung Cancer: A 2x2 Factorial Randomized Controlled Trial
Brief Title: Dexamethasone, Flurbiprofen Axetil and Delirium After Lung Cancer Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Protocol violation occurred frequently during the postoperative period.
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017[1359]-1
Record Dates: First submitted 2017-06-25; First posted 2017-06-27 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Surgery--Complications; Dexamethasone; Flubiprofen Axetil; Delirium
Keywords: Carcinoma, Non-Small-Cell Lung; Surgery; Dexamethasone; Flubiprofen Axetil; Delirium
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Delirium | interventions — Dexamethasone; dexamethasone 21-phosphate; Saline Solution; flurbiprofen axetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dexamethasone and flurbiprofen axetil (Experimental): 1. Dexamethasone 10 mg is administered before anesthesia induction.
  2. Flurbiprofen axetil 50 mg is administered before the start of surgery. Postoperative analgesia is provided with a patient-controlled analgesia pump, which is established with 100 ml of 1.25 μg/ml sufentanil and 2 mg/ml flurbiprofen axetil, programmed to deliver a 2 ml bolus with a lockout interval of 6-8 min and a background infusion of 1 ml/h.
  Interventions: Drug: Dexamethasone; Drug: Flurbiprofen axetil
- Dexamethasone and lipid microsphere (Experimental): 1. Dexamethasone 10 mg is administered before anesthesia induction.
  2. Lipid microsphere 5 ml is administered before the start of surgery. Postoperative analgesia is provided with a patient-controlled analgesia pump, which is established with 100 ml of 1.25 μg/ml sufentanil and 20 ml lipid microsphere, programmed to deliver a 2 ml bolus with a lockout interval of 6-8 min and a background infusion of 1 ml/h.
  Interventions: Drug: Dexamethasone; Drug: Lipid microsphere
- Normal saline and flurbiprofen axetil (Experimental): 1. Normal saline 2 ml is administered before anesthesia induction.
  2. Flurbiprofen axetil 50 mg is administered before the start of surgery. Postoperative analgesia is provided with a patient-controlled analgesia pump, which is established with 100 ml of 1.25 μg/ml sufentanil and 2 mg/ml flurbiprofen axetil, programmed to deliver a 2 ml bolus with a lockout interval of 6-8 min and a background infusion of 1 ml/h.
  Interventions: Drug: Normal saline; Drug: Flurbiprofen axetil
- Normal saline and lipid microsphere (Experimental): 1. Normal saline 2 ml is administered before anesthesia induction.
  2. Lipid microsphere 5 ml is administered before the start of surgery. Postoperative analgesia is provided with a patient-controlled analgesia pump, which is established with 100 ml of 1.25 μg sufentanil and 20 ml lipid microsphere, programmed to deliver a 2 ml bolus with a lockout interval of 6-8 min and a background infusion of 1 ml/h.
  Interventions: Drug: Normal saline; Drug: Lipid microsphere

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 10 mg is administered before anesthesia induction.
  Other Names: Dexamethasone sodium phosphate injection
  Arms: Dexamethasone and flurbiprofen axetil; Dexamethasone and lipid microsphere
Drug: Normal saline — Normal saline 2 ml is administered before anesthesia induction.
  Arms: Normal saline and flurbiprofen axetil; Normal saline and lipid microsphere
Drug: Flurbiprofen axetil — Flurbiprofen axetil 50 mg is administered before the start of surgery. Postoperative analgesia is provided with a patient-controlled analgesia pump, which is established with 100 ml of 1.25 μg/ml sufentanil and 2 mg/ml flurbiprofen axetil, programmed to deliver a 2 ml bolus with a lockout interval of 6-8 min and a background infusion of 1 ml/h.
  Other Names: Flurbiprofen axetil injection
  Arms: Dexamethasone and flurbiprofen axetil; Normal saline and flurbiprofen axetil
Drug: Lipid microsphere — Lipid microsphere 5 ml is administered before the start of surgery. Postoperative analgesia is provided with a patient-controlled analgesia pump, which is established with 100 ml of 1.25 μg/ml sufentanil and 20 ml lipid microsphere, programmed to deliver a 2 ml bolus with a lockout interval of 6-8 min and a background infusion of 1 ml/h.
  Other Names: Lipid microsphere injection
  Arms: Dexamethasone and lipid microsphere; Normal saline and lipid microsphere

SUMMARY:
Delirium is a common complication in elderly patients after surgery. And its occurrence is associated with worse outcomes. The causes of delirium are multifactorial but may include pain, stress response and inflammation. Dexamethasone is commonly used to prevent the occurrence of postoperative nausea and vomiting. In a randomized controlled trial, small-dose dexamethasone (8 mg) administered before anesthesia induction improved the quality of recovery in patients after cardiac surgery. Flurbiprofen axetil is commonly used to improve postoperative analgesia while decreasing the requirement of opioids. In a randomized trial of the investigators, combined use of flurbiprofen axetil with sufentanil for postoperative analgesia reduced delirium in elderly patients after orthopedic surgery. The purpose of this 2 plus 2 factorial randomized controlled trial is to test the hypothesis that combined use of dexamethasone and flurbiprofen axetil may reduce delirium in elderly patients after lung cancer surgery.

DETAILED DESCRIPTION:
Delirium is an acutely occurred, transient and fluctuating central nervous system dysfunction which is characterized by cognitive dysfunction, decreased level of consciousness, decentralized attention, and/or disturbed perception. It is a common complication in elderly patients after surgery. Systematic reviews showed that 5% to 54.4% of patients developed delirium after noncardiac surgery, and the incidences increase with age.

The development of postoperative delirium is associated with worse outcomes. For example, patients with delirium had increased postoperative complications, prolonged hospital stay, and increased in-hospital mortality; they also had worse long-term outcomes, including declined cognitive function, decreased quality of life, and increased post-hospital mortality.

The causes of delirium are multifactorial and may include pain, stress response and inflammation. Studies showed that postoperative pain is an important risk factor of delirium, whereas good postoperative analgesia reduces the incidence of delirium. Furthermore, the studies found that surgery related inflammatory response also plays an important role in the development of delirium. However, measures that can effectively prevent the occurrence of postoperative delirium are still lacking.

Dexamethasone is commonly used to prevent the occurrence of postoperative nausea and vomiting. In a randomized controlled trial, small-dose dexamethasone (8 mg) administered before anesthesia induction improved the quality of recovery in patients after cardiac surgery. Flurbiprofen axetil is commonly used to improve postoperative analgesia while decreasing the requirement of opioids. In a randomized trial of the investigators, combined use of flurbiprofen axetil with sufentanil for postoperative analgesia reduced delirium in elderly patients after orthopedic surgery.

The purpose of this 2 plus 2 factorial randomized controlled trial is to test the hypothesis that combined use of dexamethasone and flurbiprofen axetil may reduce delirium in elderly patients after lung cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 85 years old;
2. Diagnose as non-small-cell lung cancer (stage IA-IIIA);
3. Plan to undergo surgical resection;
4. Provide written informed consents.

Exclusion Criteria:

1. Clinical evidences suggest remote metastasis of the primary cancer; have received radiotherapy, chemotherapy or targeted therapy before surgery; have received previous surgery for lung cancer; diagnosed with other cancer (other than lung cancer) currently or previously;
2. History of therapy with glucocorticoids or immunosuppressants within 1 year, or therapy with non-steroidal anti-inflammatory drugs (NSAIDs) within 1 month;
3. Allergy to glucocorticoids or NSAIDs;
4. Contraindications to dexamethasone or flurbiprofen axetil, such as asthma or hives urticaria induced by aspirin or other NSAIDs; active digestive tract ulcer or bleeding, or history of repeated digestive tract ulcer or bleeding; coagulopathy (platelet count < 50*10^9/L, International Normalized Ratio > 1.4, or activated partial thromboplastin time > 4 seconds above upper limit); current therapy with lomefloxacin, norfloxacin, or enoxacin; severe cardiac dysfunction (New York heart association class 3 or above, or Left Ventricular Ejection Fraction less than 30%) or myocardial infarction within 3 months; liver injury (transaminase higher than 2 times of upper limit); kidney injury (creatinine higher than 1.5 times of upper limit); uncontrolled severe hypertension before surgery (> 180/120 mmHg);
5. American Society of Anesthesiologists (ASA) physical status class IV or higher;
6. Refuse to use patient-controlled analgesia pump after surgery;
7. Other conditions that are considered unsuitable for study participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium during the first five postoperative days. | From postoperative day 1 to postoperative day 5.
  Delirium is assessed twice daily with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU).

SECONDARY OUTCOMES:
Daily prevalence of delirium during the first five days after surgery. | From postoperative day 1 to postoperative day 5.
  Delirium is assessed twice daily with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU).
Length of stay in hospital after surgery. | From end of surgery until hospital discharge or 30 days after surgery.
  Length of stay in hospital after surgery.
Incidence of postoperative complications within 30 days after surgery. | From end of surgery until 30 days after surgery.
  Incidence of postoperative complications within 30 days after surgery.
All-cause mortality within 30 days after surgery. | From end of surgery until 30 days after surgery.
  All-cause mortality within 30 days after surgery.
Cognitive function at 30 days after surgery. | At 30 days after surgery.
  Cognitive function is assessed with Telephone Interview for Cognitive Status-Modified (TICS-m)
Quality of life at 30 days after surgery. | At 30 days after surgery.
  Quality of life is assessed with the World Health Organization Quality of Life-short version (WHOQOL-Bref).

OTHER OUTCOMES:
Richmond agitation sedation scale. | From postoperative day 1 to postoperative day 5.
  Assessed with Richmond agitation sedation scale twice daily.
Severity of pain. | From postoperative day 1 to postoperative day 5.
  Assessed twice daily with Numeric Rating Scale (NRS, an 11-score scale where 0 = no pain and 10 = the worst pain.
Cumulative analgesics consumption. | Until postoperative day 3.
  Cumulative analgesics consumption at different timepoints after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-xin Wang, Wang, Principal Investigator — Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scholz AF, Oldroyd C, McCarthy K, Quinn TJ, Hewitt J. Systematic review and meta-analysis of risk factors for postoperative delirium among older patients undergoing gastrointestinal surgery. Br J Surg. 2016 Jan;103(2):e21-8. doi: 10.1002/bjs.10062. Epub 2015 Dec 16. PMID 26676760
- [Background] Ben-David B. Anaesthesia in Cancer Surgery: Can it Affect Cancer Survival? Curr Clin Pharmacol. 2016;11(1):4-20. doi: 10.2174/1574884711666160122093154. PMID 26638975
- [Background] Bin Abd Razak HR, Yung WY. Postoperative Delirium in Patients Undergoing Total Joint Arthroplasty: A Systematic Review. J Arthroplasty. 2015 Aug;30(8):1414-7. doi: 10.1016/j.arth.2015.03.012. Epub 2015 Mar 14. PMID 25818653
- [Background] Murphy GS, Sherwani SS, Szokol JW, Avram MJ, Greenberg SB, Patel KM, Wade LD, Vaughn J, Gray J. Small-dose dexamethasone improves quality of recovery scores after elective cardiac surgery: a randomized, double-blind, placebo-controlled study. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):950-60. doi: 10.1053/j.jvca.2011.03.002. Epub 2011 May 11. PMID 21565530
- [Background] Roberts B, Rickard CM, Rajbhandari D, Turner G, Clarke J, Hill D, Tauschke C, Chaboyer W, Parsons R. Multicentre study of delirium in ICU patients using a simple screening tool. Aust Crit Care. 2005 Feb;18(1):6, 8-9, 11-4 passim. doi: 10.1016/s1036-7314(05)80019-0. PMID 18038529
- [Background] Balas MC, Happ MB, Yang W, Chelluri L, Richmond T. Outcomes Associated With Delirium in Older Patients in Surgical ICUs. Chest. 2009 Jan;135(1):18-25. doi: 10.1378/chest.08-1456. Epub 2008 Nov 18. PMID 19017895
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Ansaloni L, Catena F, Chattat R, Fortuna D, Franceschi C, Mascitti P, Melotti RM. Risk factors and incidence of postoperative delirium in elderly patients after elective and emergency surgery. Br J Surg. 2010 Feb;97(2):273-80. doi: 10.1002/bjs.6843. PMID 20069607
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Vaurio LE, Sands LP, Wang Y, Mullen EA, Leung JM. Postoperative delirium: the importance of pain and pain management. Anesth Analg. 2006 Apr;102(4):1267-73. doi: 10.1213/01.ane.0000199156.59226.af. PMID 16551935
- [Background] Halaszynski TM. Pain management in the elderly and cognitively impaired patient: the role of regional anesthesia and analgesia. Curr Opin Anaesthesiol. 2009 Oct;22(5):594-9. doi: 10.1097/ACO.0b013e32833020dc. PMID 19623056
- [Background] Rudolph JL, Ramlawi B, Kuchel GA, McElhaney JE, Xie D, Sellke FW, Khabbaz K, Levkoff SE, Marcantonio ER. Chemokines are associated with delirium after cardiac surgery. J Gerontol A Biol Sci Med Sci. 2008 Feb;63(2):184-9. doi: 10.1093/gerona/63.2.184. PMID 18314455